CLINICAL TRIAL: NCT05135273
Title: Phase 1, Dose-Escalating, Double-Blind, Randomized, Comparator-Controlled Trial of the Safety, Tolerability, and Immunogenicity of the Transmission-Blocking Vaccine Pfs230D1-EPA/Matrix-M™ Against Plasmodium Falciparum in Adults in Mali
Brief Title: Study of the Transmission-Blocking Vaccine Pfs230D1-EPA/Matrix-M Against Malaria in Adults in Mali
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Novavax (Industry); Malaria Research and Training Center, Bamako, Mali (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N°2021/210/CE/USTTB; 000576 (Other: NIH)
Record Dates: First submitted 2021-11-17; First posted 2021-11-26 (Actual); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Malaria,Falciparum
Keywords: Malaria; Reactogenicity; Antibody; Mosquito; Vaccine
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- 1a (Pilot Group) (Experimental): (n=5) to receive 12.5 µg Pfs230D1-EPA/25 µg Matrix-M on D1, D29, D57
  Interventions: Biological: Pfs230D1-EPA/Matrix-M Vaccine
- 1b (Pilot Group) (Experimental): (n=5) to receive 20 µg Pfs230D1-EPA/50 µg Matrix-M on D1, D29, D57
  Interventions: Biological: Pfs230D1-EPA/Matrix-M Vaccine
- 1c (Pilot Group) (Experimental): (n=5) to receive 40 µg Pfs230D1-EPA/50 µg Matrix-M on D1, D29, D57
  Interventions: Biological: Pfs230D1-EPA/Matrix-M Vaccine
- 1d (Pilot Group) (Active Comparator): (n=4) to receive rabies vaccine (standard dose) on D1, D29, D57
  Interventions: Biological: Verorab Rabies Vaccine
- 2a (Main Group) (Experimental): (n=15) to receive 12.5 µg Pfs230D1-EPA/25 µg Matrix-M on D1, D29, D57
  Interventions: Biological: Pfs230D1-EPA/Matrix-M Vaccine
- 2b (Main Group) (Experimental): (n=15) to receive 20 µg Pfs230D1-EPA/50 µg Matrix-M on D1, D29, D57
  Interventions: Biological: Pfs230D1-EPA/Matrix-M Vaccine
- 2c (Main Group) (Experimental): (n=15) to receive 40 µg Pfs230D1-EPA/50 µg Matrix-M on D1, D29, D57
  Interventions: Biological: Pfs230D1-EPA/Matrix-M Vaccine
- 2d (Main Group) (Active Comparator): (n=16) to receive rabies vaccine (standard dose) on D1, D29, D57
  Interventions: Biological: Verorab Rabies Vaccine

INTERVENTIONS:
Biological: Pfs230D1-EPA/Matrix-M Vaccine — Each single-use vial of Pfs230D1M-EPA contains 160 µg/mL of conjugated Pfs230D1M and 124 µg/mL or 143 µg/mL of conjugated EPA in 4 mM phosphate-buffered saline (PBS), in a volume of 0.5 mL. Each vial of Matrix-M1 contains saponin content of 0.375 mg/mL in PBS, at a pH of 7.2, in a final volume of 0.75 mL. Components will be combined in volumes defined in the protocol at point of use.
  Arms: 1a (Pilot Group); 1b (Pilot Group); 1c (Pilot Group); 2a (Main Group); 2b (Main Group); 2c (Main Group)
Biological: Verorab Rabies Vaccine — Verorab Rabies Vaccine is a purified inactivated rabies vaccine (Wistar rabies PM/WI 38 1503-3M strain) prepared on Vero cells. It is supplied as a powder and solvent for suspension for injection in a prefilled syringe. Before reconstitution, the powder is a white and homogeneous pellet. The solvent is a limpid solution.
  Arms: 1d (Pilot Group); 2d (Main Group)

SUMMARY:
Background:

Researchers are trying to develop a vaccine that will safely reduce the spread of malaria in the community by preventing mosquitos from carrying malaria from person to person.

Objective:

To assess in African adults the safety of and immune response to the administration of Pfs230D1-EPA/Matrix-M vaccine as compared to the rabies vaccine control.

Eligibility:

Healthy adults (18 to 50 years of age) who reside in Sotuba and surrounding villages in Mali

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Blood, urine, and heart tests
* Malaria comprehension exam

Participants will be randomly assigned to get either the experimental vaccine or the approved rabies vaccine. They will not know which they are getting.

Participants will get 3 doses of the study or comparator vaccine via injection in the upper arm. This occurs at the first visit, 1 month, and 2 months later.

Participants will have up to 23 scheduled visits over 14 to 16 months. Each visit includes a physical exam, and blood will be collected at most visits.

Participants will be followed up to 1 year after the final vaccination.

If participants develop an injection site rash or reaction, photographs may be taken of the site.

DETAILED DESCRIPTION:
A vaccine to interrupt malaria transmission (VIMT), targeting disruption of parasite transmission through both human and mosquito, would be a valuable additional resource in the fight to eliminate this disease. Transmission-blocking vaccines (TBVs) induce anti-sporogonic antibodies that disrupt parasite transmission to the mosquito, thereby halting transmission to another human host. Malaria-exposed populations acquire antibody against Pfs230, a parasite protein expressed by gametocytes in the human stage of P. falciparum and a surface antigen of gametes and zygotes in the mosquito stage, which suggests that a Pfs230-based vaccine may be boosted by natural malaria infection. Pfs230D1 has become one of the leading transmission-blocking antigens for consideration as a licensed TBV to be used either alone or in combination with other transmission-blocking antigens. Clinical trials with this antigen adjuvanted with either Alhydrogel or AS01 have provided very encouraging results.

This is a Phase 1, dose-escalating, randomized, double-blind, comparator-controlled study to assess the safety, tolerability, immunogenicity and transmission-blocking activity (TBA) of a 3 dose regimen of Pfs230D1-EPA/Matrix-M versus rabies vaccine in healthy adults. This will be a first-in-human assessment of Pfs230D1-EPA/Matrix-M and will be conducted as a dose-escalation trial. Participants will be randomized to 1 of the study arms to receive 1 of 3 dose levels of Pfs230D1-EPA/Matrix-M or a standard dose of comparator rabies vaccine administered as an intramuscular injection at 3 timepoints. For the 3 Pfs230D1-EPA/Matrix-M antigen dosages, we will start with a Pilot Group of 5 subjects in each Pfs230D1-EPA/Matrix-M arm and the rabies vaccine control arm. For the Pilot Group, the different dosage administrations are separated by approximately 2 weeks.

Safety outcomes will include the frequency of systemic and local adverse events and serious adverse events. Immunogenicity outcomes will be antibody responses measured by ELISA against Pfs230D1. Functional activity will be assessed by standard membrane feeding assays.

ELIGIBILITY:
INCLUSION CRITERIA:

All of the following criteria must be fulfilled for a volunteer to participate in this trial:

1. Age: > 18 years old and < 50 years old.
2. Available for the duration of the trial.
3. Known resident or long-term resident (more than 1 year) of Sotuba, Mali or surrounding villages.
4. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
5. In good general health and without clinically significant medical history in the opinion of the investigator.
6. Females of childbearing potential must be willing to use reliable contraception from 21 days prior to Study Day 0 and until 1 month after the last vaccination.

   1. A reliable method of birth control includes one of the following:

      * Confirmed pharmacologic contraceptives (parenteral) delivery.
      * Intrauterine or implantable device.
   2. EXCEPTIONS to required pregnancy prevention includes the following:

      * Postmenopausal state: defined as no menses for 12 months without an alternative medical cause.
      * Surgical sterilization.
7. Willing to have blood samples stored for future research.

EXCLUSION CRITERIA:

An individual will be excluded from participating in this trial if any one of the following criteria is fulfilled:

1. Pregnant, as determined by a positive urine or serum beta human choriogonadotropin (β hCG) test (if female). NOTE: Pregnancy is also a criterion for discontinuation of any further vaccine dosing.
2. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and comply with the study protocol at a level appropriate for the subject's age.
3. Hemoglobin, white blood cell (WBC), absolute neutrophil count, or platelet levels outside the local laboratory-defined limits of normal. (Subjects may be included at the investigator's discretion for "not clinically significant" values outside of normal range and ≤ Grade 2.)
4. Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of normal. (Subjects may be included at the investigator's discretion for "not clinically significant" values outside of normal range and ≤ Grade 2.)
5. Infected with HIV.
6. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies.
7. History of receiving any investigational product within the past 30 days.
8. Current or planned participation in an investigational vaccine study until the time period of the last required study visit under this protocol.
9. Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
10. History of a severe allergic reaction or anaphylaxis.
11. Known:

    * Severe asthma, defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past 2 years, or that has required the use of oral or parenteral corticosteroids at any time during the past 2 years.
    * Autoimmune or antibody-mediated disease including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjögren's syndrome, or autoimmune thrombocytopenia.
    * Immunodeficiency syndrome.
    * Seizure disorder (exception: history of simple febrile seizures).
    * Asplenia or functional asplenia.
    * Use of chronic (≥14 days) oral or intravenous (IV) corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of Study Day 0.
    * Allergy to latex or neomycin.
12. Receipt of:

    * Live vaccine within 4 weeks prior to enrollment or a killed vaccine within 2 weeks prior to enrollment.
    * Immunoglobulins and/or blood products within the past 6 months.
    * Investigational malaria vaccine in the last 2 years.
13. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial, interfere with the evaluation of the study objectives, or would render the subject unable to comply with the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Duffy, MD, Study Chair — National Institute of Allergy and Infectious Diseases (NIAID); Issaka Sagara, MD, Principal Investigator — Malaria Research and Training Center, Bamako, Mali
Locations (1):
- Malaria Research Training Center, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coelho CH, Tang WK, Burkhardt M, Galson JD, Muratova O, Salinas ND, Alves E Silva TL, Reiter K, MacDonald NJ, Nguyen V, Herrera R, Shimp R, Narum DL, Byrne-Steele M, Pan W, Hou X, Brown B, Eisenhower M, Han J, Jenkins BJ, Doritchamou JYA, Smelkinson MG, Vega-Rodriguez J, Truck J, Taylor JJ, Sagara I, Healy SA, Renn JP, Tolia NH, Duffy PE. A human monoclonal antibody blocks malaria transmission and defines a highly conserved neutralizing epitope on gametes. Nat Commun. 2021 Mar 19;12(1):1750. doi: 10.1038/s41467-021-21955-1. PMID 33741942
- [Background] Datoo MS, Natama MH, Some A, Traore O, Rouamba T, Bellamy D, Yameogo P, Valia D, Tegneri M, Ouedraogo F, Soma R, Sawadogo S, Sorgho F, Derra K, Rouamba E, Orindi B, Ramos Lopez F, Flaxman A, Cappuccini F, Kailath R, Elias S, Mukhopadhyay E, Noe A, Cairns M, Lawrie A, Roberts R, Valea I, Sorgho H, Williams N, Glenn G, Fries L, Reimer J, Ewer KJ, Shaligram U, Hill AVS, Tinto H. Efficacy of a low-dose candidate malaria vaccine, R21 in adjuvant Matrix-M, with seasonal administration to children in Burkina Faso: a randomised controlled trial. Lancet. 2021 May 15;397(10287):1809-1818. doi: 10.1016/S0140-6736(21)00943-0. Epub 2021 May 5. PMID 33964223
- [Background] Healy SA, Anderson C, Swihart BJ, Mwakingwe A, Gabriel EE, Decederfelt H, Hobbs CV, Rausch KM, Zhu D, Muratova O, Herrera R, Scaria PV, MacDonald NJ, Lambert LE, Zaidi I, Coelho CH, Renn JP, Wu Y, Narum DL, Duffy PE. Pfs230 yields higher malaria transmission-blocking vaccine activity than Pfs25 in humans but not mice. J Clin Invest. 2021 Apr 1;131(7):e146221. doi: 10.1172/JCI146221. PMID 33561016
- [Derived] Cao Y, da Silva Araujo M, Lorang CG, Dos Santos NAC, Tripathi A, Vinetz J, Kumar N. Distinct immunogenicity outcomes of DNA vaccines encoding malaria transmission-blocking vaccine target antigens Pfs230D1M and Pvs230D1. Vaccine. 2025 Feb 15;47:126696. doi: 10.1016/j.vaccine.2024.126696. Epub 2025 Jan 8. PMID 39787798

RESULTS

PARTICIPANT FLOW:
Groups:
- 12.5 µg Dose (Arm 1a Pilot): Participants received 3 doses of 12.5 µg Pfs230D1-EPA/25 µg Matrix-M
  Pilot/safety: Dosing interval on days: 1, 29, 57
- 20 µg Dose (Arm 1b Pilot): Participants received 3 doses of 20 µg Pfs230D1-EPA/50 µg Matrix-M
  Pilot/safety: Dosing interval on days: 1, 29, 57
- 40 µg Dose (Arm 1c Pilot): Participants received 3 doses of 40 µg Pfs230D1-EPA/50 µg Matrix-M
  Pilot/safety: Dosing interval on days: 1, 29, 57
- Rabies Comparator (Arm 1d Pilot): Participants received 3 doses of rabies vaccine (standard dose)
  Pilot/safety: Dosing interval on days: 1, 29, 57
- 12.5 µg (Arm 2a Main): Participants received 3 doses of 12.5 µg Pfs230D1-EPA/25 µg Matrix-M
  Main/Safety/efficacy: Dosing interval on days: 1, 29, 57
- 20 µg Dose (Arm 2b Main): Participants received 3 doses of 20 µg Pfs230D1-EPA/50 µg Matrix-M
  Main/Safety/efficacy: Dosing interval on days: 1, 29, 57
- 40 µg Dose (Arm 2c Main): Participants received 3 doses of 40 µg Pfs230D1-EPA/50 µg Matrix-M
  Main/Safety/efficacy: Dosing interval on days: 1, 29, 57
- Rabies Comparator (Arm 2d Main): Participants received 3 doses of rabies vaccine (standard dose)
  Main/Safety/efficacy: Dosing interval on days: 1, 29, 57
Period: Overall Study
Arm/Group | 12.5 µg Dose (Arm 1a Pilot) | 20 µg Dose (Arm 1b Pilot) | 40 µg Dose (Arm 1c Pilot) | Rabies Comparator (Arm 1d Pilot) | 12.5 µg (Arm 2a Main) | 20 µg Dose (Arm 2b Main) | 40 µg Dose (Arm 2c Main) | Rabies Comparator (Arm 2d Main)
Started | 5 | 5 | 5 | 4 | 14 | 14 | 15 | 16
Completed | 5 | 5 | 5 | 4 | 13 | 13 | 14 | 15
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Not completed — Recruited into the army | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Moved away from study site | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Travel | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 12.5 µg Dose (Arm 1a Pilot) | 20 µg Dose (Arm 1b Pilot) | 40 µg Dose (Arm 1c Pilot) | Rabies Comparator (Arm 1d Pilot) | 12.5 µg (Arm 2a Main) | 20 µg Dose (Arm 2b Main) | 40 µg Dose (Arm 2c Main) | Rabies Comparator (Arm 2d Main) | Total
Number analyzed (Participants) | 5 | 5 | 5 | 4 | 14 | 14 | 15 | 16 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 4 | 14 | 14 | 15 | 16 | 78
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 3 | 6 | 4 | 4 | 5 | 29
  Male | 4 | 3 | 1 | 1 | 8 | 10 | 11 | 11 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 5 | 4 | 14 | 14 | 15 | 16 | 78
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mali | 5 | 5 | 5 | 4 | 14 | 14 | 15 | 16 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Local and Systemic Adverse Events (AEs) to Assess the Safety of the Study Drug
Description: The analyses included only subjects who received at least one vaccination
Time Frame: Adverse Events monitored/assessed for 7 days after each vaccination at days 1, 29, and 57; All-Cause Mortality monitored/assessed through 14 months
Measure: Number; unit: Adverse Events
Arm/Group | 12.5 µg Dose (Arm 1a Pilot) | 20 µg Dose (Arm 1b Pilot) | 40 µg Dose (Arm 1c Pilot) | Rabies Comparator (Arm 1d Pilot) | 12.5 µg (Arm 2a Main) | 20 µg Dose (Arm 2b Main) | 40 µg Dose (Arm 2c Main) | Rabies Comparator (Arm 2d Main)
Number analyzed (Participants) | 5 | 5 | 5 | 4 | 14 | 14 | 15 | 16
Adverse Events | 34 | 24 | 23 | 16 | 45 | 60 | 58 | 39

2. Primary Outcome: Number of Local and Systemic Serious Adverse Events (SAEs) to Assess the Safety of the Study Drug
Time Frame: Serious Adverse Events monitored/assessed for 7 days after each vaccination at days 1, 29, and 57; All-Cause Mortality monitored/assessed through 14 months
Measure: Number; unit: Serious Adverse Events
Arm/Group | 12.5 µg Dose (Arm 1a Pilot) | 20 µg Dose (Arm 1b Pilot) | 40 µg Dose (Arm 1c Pilot) | Rabies Comparator (Arm 1d Pilot) | 12.5 µg (Arm 2a Main) | 20 µg Dose (Arm 2b Main) | 40 µg Dose (Arm 2c Main) | Rabies Comparator (Arm 2d Main)
Number analyzed (Participants) | 5 | 5 | 5 | 4 | 14 | 14 | 15 | 16
Serious Adverse Events | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed for 7 days after each vaccination at days 1, 29, and 57; All-Cause Mortality monitored/assessed through 14 months
Arm/Group | 12.5 µg Dose (Arm 1a Pilot) | 20 µg Dose (Arm 1b Pilot) | 40 µg Dose (Arm 1c Pilot) | Rabies Comparator (Arm 1d Pilot) | 12.5 µg (Arm 2a Main) | 20 µg Dose (Arm 2b Main) | 40 µg Dose (Arm 2c Main) | Rabies Comparator (Arm 2d Main)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/4 | 0/14 | 0/14 | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/5 | 0/5 | 0/4 | 0/14 | 0/14 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 5/5 | 4/4 | 12/14 | 14/14 | 15/15 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12.5 µg Dose (Arm 1a Pilot) (N=5) | 20 µg Dose (Arm 1b Pilot) (N=5) | 40 µg Dose (Arm 1c Pilot) (N=5) | Rabies Comparator (Arm 1d Pilot) (N=4) | 12.5 µg (Arm 2a Main) (N=14) | 20 µg Dose (Arm 2b Main) (N=14) | 40 µg Dose (Arm 2c Main) (N=15) | Rabies Comparator (Arm 2d Main) (N=16)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12.5 µg Dose (Arm 1a Pilot) (N=5) | 20 µg Dose (Arm 1b Pilot) (N=5) | 40 µg Dose (Arm 1c Pilot) (N=5) | Rabies Comparator (Arm 1d Pilot) (N=4) | 12.5 µg (Arm 2a Main) (N=14) | 20 µg Dose (Arm 2b Main) (N=14) | 40 µg Dose (Arm 2c Main) (N=15) | Rabies Comparator (Arm 2d Main) (N=16)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Candidiasis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Decreased appetite (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysentery (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear infection (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (2)
Headache (General disorders) | 3 (4) | 0 (0) | 3 (4) | 0 (0) | 4 (6) | 3 (4) | 10 (16) | 4 (5)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 3 (6) | 3 (6) | 0 (0) | 7 (9) | 9 (11) | 10 (12) | 1 (1)
Leuokocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 3 (3) | 3 (4) | 1 (1) | 2 (4) | 4 (7) | 3 (5) | 3 (4) | 5 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 1 (2) | 1 (1) | 1 (1) | 1 (2) | 5 (9) | 0 (0) | 3 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parasitic gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (3) | 1 (2) | 2 (3) | 3 (3) | 9 (10) | 5 (6) | 8 (10)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinobronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 1 (1)
Tonsillitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT05135273/Prot_SAP_000.pdf